CLINICAL TRIAL: NCT00129298
Title: Tiagabine for the Treatment of Cocaine Dependence in Methadone-Maintained Individuals
Brief Title: Effectiveness of Tiagabine for Cocaine Dependence in Methadone-Maintained Individuals - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Gerardo Gonzalez, MD, Yale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NIDA-17782-1; R01-17782-1; DPMC
Record Dates: First submitted 2005-08-04; First posted 2005-08-11 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2007-12

CONDITIONS: Cocaine-Related Disorders; Opiate Dependence
Keywords: cocaine abuse; opiate dependent; tiagabine; methadone
MeSH Terms: conditions — Cocaine-Related Disorders; Opioid-Related Disorders | interventions — Tiagabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Tiagabine
  Interventions: Drug: Tiagabine
- 2 (Placebo Comparator): Matching placebo
  Interventions: Drug: Tiagabine

INTERVENTIONS:
Drug: Tiagabine — The tiagabine group will start receiving tiagabine 4mg in the evening of the first day on week 2. The dose will be titrated every third day, until the target dose of 32mg/day is achieved by week 5. The study medication must be titrated to 32 mg/day or to the subject's maximum tolerated dose (MTD).
  Other Names: Gabatril

SUMMARY:
Many opioid-dependent individuals are also dependent on cocaine. Methadone is a widely used and effective method for treating opioid dependence. However, it is not effective in treating other drugs of abuse. The purpose of this study is to determine the effectiveness of another drug, tiagabine, for treating cocaine dependence in opioid-dependent individuals already receiving methadone treatment.

DETAILED DESCRIPTION:
For over 30 years, methadone has been used to treat opioid addiction. Since methadone is effective in reducing withdrawal symptoms, it is used as a method of detoxification for opiate addicts. However, methadone is not effective in treating other drugs of abuse, such as cocaine. Tiagabine is a drug that enhances levels of gamma aminobutyric acid (GABA), a chemical found in the brain and spinal cord. The objective of this study is to determine the effectiveness of tiagabine in modifying cocaine-using behavior and reducing opiate withdrawal symptoms among newly admitted methadone-treated patients.

This 16-week, double-blind, placebo-controlled clinical trial will involve 120 participants who are both cocaine- and opioid- dependent. Participants will be randomly assigned to receive either tiagabine or placebo, while concurrently receiving methadone treatment. Baseline cocaine use will be determined during the first two weeks of treatment. The study will include three overlapping phases. The first phase will include a one-week fixed methadone induction (Week 1), as well as flexible methadone stabilization (Weeks 2-13). Phase two will consist of a 12-week treatment period (Weeks 2-13). This will consist of tiagabine induction and stabilization. Phase three will include a 4-week taper, detoxification, or transfer period (Weeks 14-17). After completion of treatment, a 3-month follow-up visit will occur.

ELIGIBILITY:
Inclusion Criteria:

* Currently not enrolled in methadone-maintenance treatment
* Demonstration of current opioid dependence as determined by the study physician, a self-reported history of opioid dependence for one year, and a positive urine test for opiates
* Current cocaine abuser with self-reported use of cocaine at least 1 time each week within the month prior to study entry, positive urine screen for cocaine, and score greater than 3 on the Severity Dependence Scale
* Women of childbearing age are eligible under the following conditions: negative pregnancy test at initial screening, adequate contraceptive use throughout the study, monthly pregnancy tests, and acknowledgement of fetal toxicity risks due to medication

Exclusion Criteria:

* Current diagnosis of other drug or alcohol dependence (other than opiates, cocaine, or tobacco)
* Serious medical illness (e.g., major heart, kidney, endocrine, or liver disease, or serious neurological disorders, including history of seizures)
* Current diagnosis of a serious psychiatric illness or history of psychosis, schizophrenia, or bipolar type I disorder
* Suicidal or homicidal thoughts
* Currently taking psychotropic medications
* Women who are pregnant, nursing, refuse to use a reliable form of contraception, or refuse monthly pregnancy testing
* Greater than 3 times the normal level in liver screening function test (SGOT or SGPT)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2004-12; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Thrice weekly Urine toxicology | 13 weeks

SECONDARY OUTCOMES:
Self reports of cocaine and opioid use. | 13 weeks
Opioid withdrawal symptoms | 13 weeks
Adverse events | 13 weeks
cocaine craving | 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo Gonzalez, M.D., Principal Investigator — Yale University